CLINICAL TRIAL: NCT06541704
Title: A Multicenter, Randomized, Double-Masked, Placebo-Controlled Phase 3 Study of the Efficacy, Safety, and Tolerability of Subcutaneously Administered Pozelimab in Combination With Cemdisiran or Cemdisiran Alone in Participants With Geographic Atrophy Secondary to Age-Related Macular Degeneration
Brief Title: A Study Investigating Subcutaneously Administered Pozelimab in Combination With Cemdisiran or Cemdisiran Alone in Adult Participants With Geographic Atrophy
Acronym: SIENNA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R3918-AMD-2326; 2023-509547-27-00 (EU CTIS Number)
Record Dates: First submitted 2024-08-02; First posted 2024-08-07 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Age-related Macular Degeneration (AMD); Geographic Atrophy (GA)
Keywords: GA secondary to AMD
MeSH Terms: conditions — Macular Degeneration; Geographic Atrophy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Pozelimab + Cemdisiran treatment group (Experimental): Randomized 1:1:1
  Interventions: Drug: Pozelimab; Drug: Cemdisiran
- Cemdisiran monotherapy treatment group (Experimental): Randomized 1:1:1
  Interventions: Drug: Cemdisiran
- Placebo treatment group (Placebo Comparator): Randomized 1:1:1
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pozelimab — Subcutaneous (SC) injection
  Other Names: REGN3918
  Arms: Pozelimab + Cemdisiran treatment group
Drug: Cemdisiran — SC injection
  Other Names: ALN-CC5
  Arms: Cemdisiran monotherapy treatment group; Pozelimab + Cemdisiran treatment group
Drug: Placebo — SC injection
  Arms: Placebo treatment group

SUMMARY:
This study is researching experimental (study) drugs called pozelimab and cemdisiran. The study is focused on participants who have Geographic Atrophy (GA) caused by Age-related Macular Degeneration (AMD). Geographic atrophy is a medical term that refers to later-stage cases of AMD which is an eye condition affecting central vision (what one sees straight ahead).

The purpose of this study is to evaluate the progression rate of Geographic Atrophy in eyes of patients treated with cemdisiran alone or in combination with pozelimab compared to those treated with placebo.

The study is looking at several other research questions, including:

* What side effects may happen from taking the study drug(s)
* How much study drug(s) are in the blood at different times
* Whether the body makes antibodies against the study drug(s) (which could make the study drug(s) less effective or could lead to side effects)

ELIGIBILITY:
Key Inclusion Criteria:

1. Study eye with diagnosis of GA of the macula secondary to AMD as described in the protocol
2. Total GA area in the study eye measuring between ≥2.5 mm^2 and ≤17.5 mm^2 as described in the protocol
3. BCVA of 55 letters or better using ETDRS charts (20/80 Snellen equivalent) in the study eye as described in the protocol
4. Sufficiently clear ocular media, adequate pupillary dilation and fixation to permit quality fundus imaging in the study eye as described in the protocol
5. Willing and able to comply with clinic visits and study-related procedures, including completion of the full series of meningococcal vaccinations and pneumococcal vaccination required per protocol

Key Exclusion Criteria:

1. GA in either eye due to causes other than AMD, such as Stargardt disease, cone rod dystrophy or toxic maculopathies like hydroxychloroquine maculopathy
2. History or current evidence of Macular Neovascularization (MNV) and/or exudation or Peripapillary Choroidal Neovascularization (PPCNV) in either eye as described in the protocol
3. Prior or current Intravitreal (IVT) treatment of any kind for any indication in study eye or fellow eye, except approved or investigational IVT complement inhibitor therapy or anti-VEGF therapy, as long as last dose was ≥6 months prior to randomization
4. Prior intraocular surgery except cataract extraction or minimally invasive glaucoma surgery in study eye as long as date of these procedures was ≥3 months prior to randomization
5. Comorbid progressive ocular condition (eg, diabetic retinopathy, macular edema, uncontrolled glaucoma, full thickness macular hole) in study eye that could affect central vision and confound study
6. Any ophthalmologic condition that reduces the clarity of the media and that, in the opinion of the investigator interferes with ophthalmologic examination of the study eye (e.g., advanced cataract or corneal abnormalities) as described in the protocol

   Systemic Exclusion criteria
7. History or current use of systemic complement inhibitor therapy within 6 months prior to randomization as described in the protocol
8. History of solid organ or bone marrow transplantation
9. Use of chronic (>14 days) systemic corticosteroids (oral or parenteral, ≥20 mg oral prednisone or equivalent) within the previous 30 days prior to the first screening visit as described in the protocol
10. Current or prior use of systemic immunosuppressive therapy other than corticosteroids within 12 months prior to randomization or the likelihood of treatment with any such agent during the study inclusive of the screening period as described in the protocol
11. Not meeting meningococcal or pneumococcal vaccination requirements as described in the protocol
12. Carrier of Neisseria meningitidis based on culture collected during screening
13. Has a hemoglobin A1C ≥ 8.0% during screening as described in the protocol

NOTE: Other protocol-defined Inclusion/ Exclusion Criteria apply

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 975 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2027-11-29 (Estimated); Study Completion 2032-05-21 (Estimated)

PRIMARY OUTCOMES:
Growth rate (slope) of total GA lesion area (mm^2 /year) from baseline, measured by Fundus Autofluorescence (FAF) | To week 52

SECONDARY OUTCOMES:
Loss of Best Corrected Visual Acuity (BCVA) ≥15 letters [Early Treatment Diabetic Retinopathy Study (ETDRS)] from baseline | At week 52 and week 104
Change from baseline in Low-Contrast quantitative Visual Acuity (LC-qVA) | At week 52 and week 104
Change from baseline in Low-Luminance Low-Contrast quantitative Visual Acuity (LL-LC-qVA) | At week 52 and week 104
Change from baseline in quantitative Contrast Sensitivity Function (qCSF) | At week 52 and week 104
Growth rate (slope) of total GA lesion area (mm^2 /year) from baseline measured by FAF | To week 104
Concentrations of total pozelimab in serum | Through week 52 and through week 104
Concentrations of total cemdisiran in plasma | Through week 52 and through week 104
Change from baseline in concentration of total Complement component 5 (C5) | Through week 52 and through week 104
Incidence of Antidrug antibody (ADA) to pozelimab | Through week 52 and through week 104
Magnitude of ADA to pozelimab | Through week 52 and through week 104
Incidence of ADA to cemdisiran | Through week 52 and through week 104
Magnitude of ADA to cemdisiran | Through week 52 and through week 104
Incidence of Neutralizing Antibody (NAb) to pozelimab | Through week 52 and through week 104
Occurrence of Treatment-Emergent Adverse Events (TEAEs) | Through week 52, 104, 140 and week 296
Severity of TEAEs | Through week 52, 104, 140 and week 296

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (198):
- United States (141):
  - Barnet Dulaney Perkins Eye Center, Phoenix, Arizona
  - Associated Retina Consultants, Phoenix, Arizona
  - Retinal Research Institute, Phoenix, Arizona
  - Retina Macula Institute of Arizona, Scottsdale, Arizona
  - Retina Associates of Tuscan, Tucson, Arizona
  - Retina Partners of Northwest Arkansas, PLLC, Springdale, Arkansas
  - Retina Vitreous Associates Medical Group, Beverly Hills, California
  - Retina Specialists of Beverly Hills- Department of Ophthalmology, Beverly Hills, California
  - The Retina Partners, Encino, California
  - Eye Medical Center of Fresno, Fresno, California
  - Retina Consultants of Orange County, Fullerton, California
  - Salehi Retina Institute dba Retina Associates of Southern California, Huntington Beach, California
  - University of California Irvine, Irvine, California
  - University of California San Diego, Jacobs Retina Center, La Jolla, California
  - South Coast Retina Center, Long Beach, California
  - American Institute of Research, Los Angeles, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Retinal Consultants Medical Group Inc Modesto, Modesto, California
  - Northern California Retina Vitreous Associates Medical Group, Inc., Mountain View, California
  - California Retina Consultants, Oxnard, California
  - Desert Retina Consultants, Palm Desert, California
  - California Eye Specialists Medical Group Inc., Pasadena, California
  - Retina Consultants San Diego, Poway, California
  - California Eye Specialists Medical Group, Inc., Redlands, California
  - Optic Eye Care, Rowland Heights, California
  - UC Davis Health Eye Center, Sacramento, California
  - Vrmg Inc, Sacramento, California
  - Retinal Consultants Medical Group (RCMG) - Greenback Lane Retina Center, Sacramento, California
  - West Coast Retina Medical Group, Inc., San Francisco, California
  - Orange County Retina Medical Group, Santa Ana, California
  - Macula Retina Vitreous Research Institute, Torrance, California
  - University of Colorado, Aurora, Colorado
  - Retina Consultants of Southern Colorado, Colorado Springs, Colorado
  - Southwest Retina Research Center, Durango, Colorado
  - Colorado Retina - Lakewood, Lakewood, Colorado
  - Eye care Center of Northern Colorado doing business as Advanced Vision Research Institute, Longmont, Colorado
  - Retina Group of New England, Waterford, Connecticut
  - Retina Center Tampa Bay- Ophthalmology, Bayonet Point, Florida
  - Advanced Research, Coral Springs, Florida
  - Retina Group of Florida, Fort Lauderdale, Florida
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - Florida Retina Institute, Jacksonville Perimeter Park- Ophthalmology, Jacksonville, Florida
  - Florida Retina Consultants, Lakeland, Florida
  - Bascom Palmer Eye Institute, Naples, Florida
  - Florida Retina Institute - Orlando, Orlando, Florida
  - Retina Care Specialists, Palm Beach Gardens, Florida
  - Eye Associates of Pinellas, Pinellas Park, Florida
  - Retina Group of Florida, RAS-Sarasota Retina Center-Ophthalmology, Sarasota, Florida
  - Retina Vitreous Associates of Florida Saint Petersburg, St. Petersburg, Florida
  - University of South Florida Ophthalmology, Tampa, Florida
  - Center for Retina and Macular Disease, Winter Haven, Florida
  - Southeast Retina Center, Augusta, Georgia
  - Georgia Retina - Marietta, Marietta, Georgia
  - University of Illinois at Chicago, Chicago, Illinois
  - Retinal Vitreal Consultants, Chicago, Illinois
  - The University of Chicago, Chicago, Illinois
  - University Retina and Macula Associates PC - Lemont, Lemont, Illinois
  - Illinois Retina Associates, Oak Park, Illinois
  - Springfield Clinic Main Campus East, Springfield, Illinois
  - Retina Associates, LLC, Lenexa, Kansas
  - Retina Associates New Orleans, Metairie, Louisiana
  - Ross Davis Retina, Metairie, Louisiana
  - Ochsner Health, New Orleans, Louisiana
  - Eye Assoc. of NE LA dba Haik Humble Eye Ctr, West Monroe, Louisiana
  - Eye Associates of Northeast Louisiana dba Haik Humble Eye Center, West Monroe, Louisiana
  - The Retina Care Center, Baltimore, Maryland
  - The Retina Group of Washington, Chevy Chase, Maryland
  - Cumberland Valley Retina Consultants-Ophthalmology, Hagerstown, Maryland
  - Mid Atlantic Retina Specialist, Hagerstown, Maryland
  - Massachusetts Eye And Ear Infirmary, Boston, Massachusetts
  - Opthalmic Consultants of Boston, Boston, Massachusetts
  - New England Retina Consultants, PC, Springfield, Massachusetts
  - Mississippi Retina Associates, Madison, Mississippi
  - Deep Blue Retina Clinical Research PLLC, Southaven, Mississippi
  - Retina Research Institute, LLC, St Louis, Missouri
  - Mid Atlantic Retina - Cherry Hill, Cherry Hill, New Jersey
  - New Jersey Retina, Teaneck, New Jersey
  - New Jersey Retina, Toms River, New Jersey
  - Vision Research Center at Eye Associates of New Mexico, Albuquerque, New Mexico
  - University of New Mexico, HSC, Albuquerque, New Mexico
  - Sight MD, Brentwood, New York
  - Retina Vitreous Surgeons of Central New York, PC, Liverpool, New York
  - MaculaCare, PLLC, New York, New York
  - New York Ear & Eye- East 85th, New York, New York
  - Retina Associates of New York, Ophthalmology, New York, New York
  - Seeta Eye center, Poughkeepsie, New York
  - Western Carolina Retinal Associates, Asheville, North Carolina
  - NC Retina Associates, Cary, North Carolina
  - Graystone Eye, Hickory, North Carolina
  - North Carolina Retina Associates, Wake Forest, North Carolina
  - Piedmont Retina Specialist, Winston-Salem, North Carolina
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Midwest Retina, Inc, Dublin, Ohio
  - Retina Vitreous Center - Edmond, Edmond, Oklahoma
  - Tulsa Retina Consultants, Tulsa, Oklahoma
  - Verum Research LLC, Eugene, Oregon
  - Retina Northwest, The Highlands Building, Portland, Oregon
  - EyeHealth Northwest, Portland, Oregon
  - OHSU-Casey Eye Institute, Marquam Hill-Ophthalmology, Portland, Oregon
  - Cascade Medical Research Institute LLC, Springfield, Oregon
  - Mid Atlantic Retina, Bethlehem, Pennsylvania
  - Erie Retinal Surgery & Erie Retina Research, Erie, Pennsylvania
  - Mid Atlantic Retina, Wills Eye Hospital, Philadelphia, Pennsylvania
  - Vision Research Solutions - the Eye Institute, Philadelphia, Pennsylvania
  - Sewickley Eye Group, Sewickley, Pennsylvania
  - Retina Consultants of Carolina, Greenville, South Carolina
  - Charleston Neuroscience Institute LLC, Ladson, South Carolina
  - Charleston Neuroscience Institute, LLC, Mt. Pleasant, South Carolina
  - Palmetto Retina Center, West Columbia, South Carolina
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Tennessee Retina, PC, Nashville, Tennessee
  - Vanderbilt Eye Institute, Nashville, Tennessee
  - Retina Research Institute of Texas, Abilene, Texas
  - Austin Research Center for Retina, Austin, Texas
  - Austin Retina Associates, Austin, Texas
  - Austin Clinical Research LLC, Austin, Texas
  - Retina Consultants Texas, Bellaire, Texas
  - Star Retina PLLC, Burleson, Texas
  - Retina Foundation of the Southwest, Dallas, Texas
  - Texas Retina Associates, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Retina Consultants of Texas, Katy, Texas
  - Valley Retina Institute, P.A., McAllen, Texas
  - Red River Research Partners (Formerly AXIS Clinical), Plano, Texas
  - Austin Retina Associates, Round Rock, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Retina Associates of South Texas, San Antonio, Texas
  - Retina Consultants of Texas, San Antonio, Texas
  - Retina Consultants of Texas Brown Retina Institute, San Antonio, Texas
  - Retina Center of Texas, Southlake, Texas
  - Retina Consultants Texas, The Woodlands, Texas
  - Retina Associates Of Utah Retina Specialist, Salt Lake City, Utah
  - Rocky Mountain Retina Consultants, Salt Lake City, Utah
  - Retina Group of Washington, Fairfax, Virginia
  - Piedmont Eye Center, Lynchburg, Virginia
  - Virginia Eye Institute, Richmond, Virginia
  - Retina Institute of Virginia, Richmond, Virginia
  - Spokane Eye Clinical Research, Spokane, Washington
  - West Virginia University Eye Institute, Morgantown, West Virginia
- Austria (3):
  - Medical University Graz, Graz, Styria
  - Medical University of Vienna, Vienna
  - VIROS - Vienna Institute for Research in Ocular Surgery, Vienna
- Canada (2):
  - Retina Centre of Ottawa - Department of Ophthalmology, Ottawa, Ontario
  - Centre Hospitalier Universitaire de Quebec Universite Laval, Québec
- France (9):
  - Centre Hospitalier Universitaire de Nice, Nice, Alpes Maritimes
  - Hopital Saint Joseph, Marseille, Bouches Du Rhone
  - Centre Hospitalier Universitaire De Poitiers, Poitiers, Nouvelle-Aquitaine
  - Centre Hospitalier Intercommunal de Creteil, Créteil
  - Centre Hospitalier Universitaire Francois Mitterrand, Dijon
  - Hopital De La Croix-Rousse, Lyon
  - Centre Monticelli Paradis, Marseille
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - Hopital Lariboisiere, Paris
- Germany (11):
  - Charite - Universitaetsmedizin Berlin, Berlin, Brandenburg
  - Augenzentrum Frankfurt, Frankfurt am Main, Hesse
  - Universitaetsklinikum Marburg, Klinik fuer Augenheilkunde, Marburg, Hesse
  - Dietrich Bonhoeffer Klinikum, Neubrandenburg, Mecklenburg-Vorpommern
  - Klinik fur Augenheilkunde Universitatsklinikum Dusseldorf, Düsseldorf, North Rhine-Westphalia
  - Universitaetsklinikum Muenster, Münster, North Rhine-Westphalia
  - Saarland University Medical Center, Homburg, Saarland
  - Knappschaftsklinikum Saar GmbH- Eye Clnic Sulzbach, Sulzbach, Saarland
  - University Hospital Hamburg Eppendorf, Hamburg
  - University Medical Center of the Johannes Gutenberg-University Mainz, Mainz
  - St. Franziskus-Hospital, Münster
- Hungary (5):
  - Ganglion Medical Center, Pécs, Baranya
  - University Of Szeged, Szeged, Csongrad-Csanad
  - University Of Debrecen, Hungary, Debrecen, Hajdú-Bihar
  - Semmelweis University, Budapest
  - Budapest Retina Associates, Budapest
- Italy (8):
  - University Hospital PTV, Rome, Lazio
  - Fondazione Policlinico Gemelli, Rome, Lazio
  - IRCCS MultiMedica, Milan, Lombardy
  - Ospedale San Raffaele (HSR) - Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS), Milan, Milano
  - Azienda Ospedaliero Universitaria Careggi, Florence, Tuscany
  - Azienda Ospedaliero Universitaria delle Marche, Ancona
  - Universita degli Studi di Milano, Milan
  - Fondazione G.B.Bietti Per Lo Studio E La Ricerca In Oftalmologia, Rome
- Poland (3):
  - Oftalmika Sp. z o.o., Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Caminomed, Tarnowskie Góry, Silesian Voivodeship
  - Centrum Diagnostyki I Mikrochirurgii Oka Lens Sp zoo, Olsztyn, Warmian-Masurian Voivodeship
- Spain (10):
  - Hospital Arruzafa, Córdoba, Andalusia
  - Bellvitge University Hospital, L'Hospitalet de Llobregat, Barcelona
  - Hospital de Terrassa (Consorci Sanitari de Terrassa), Terrassa, Barcelona
  - Oftalvist Clinic. IMED Hospital, Burjassot, Valencia
  - Centro de Oftalmologia Barraquer, Barcelona
  - Instituto de Microcirugia Ocular, Barcelona
  - Institut Catala De Retina S.L., Barcelona
  - Hospital Universitario Virgen Macarena, Seville
  - Fundacion Aiken De La Comunitat Valenciana, Valencia
  - Hospital Clinico Universitario Lozano Blesa. IIS Aragon, Zaragoza
- United Kingdom (6):
  - Liverpool University Hospitals NHS Foundation Trust-Royal Liverpool University Hospital, St Paul's Eye Unit-Ophthalmology, Liverpool, Merseyside
  - York and Scarborough Teaching Hospitals NHS Foundation Trust, York, North Yorkshire
  - University Hospitals Bristol NHS Foundation Trust, Bristol
  - Moorfields Eye Hospital NHS Foundation Trust, Moorfields Eye Hospital, London
  - Imperial College Healthcare NHS Trust, London
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/